CLINICAL TRIAL: NCT00250042
Title: A Phase II Study of Gleevec and Arsenic Trioxide in Patients With CML Who Fail to Achieve a Complete Response to Initial Gleevec Treatment
Brief Title: A Phase II Study of Gleevec and Arsenic Trioxide in Patients With CML Who Fail Gleevec
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0604C
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2009-12

CONDITIONS: Leukemia, Other; Cancer
MeSH Terms: conditions — Leukemia; Neoplasms | interventions — Imatinib Mesylate; Arsenic Trioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Gleevec and Arsenic Trioxide — Pts. who fit the inclusion criteria, & were on imatinib, 400 mg/day, will be treated with a month of imatinib at 800 mg/d in divided doses (400mg bid) & then started on arsenic trioxide. Pts. already on imatinib 800 mg/day may be started on arsenic trioxide. Pts. unable to tolerate 800 mg/d should be treated at the max. dose tolerated above 400 mg/d. A total of 16 weeks of arsenic trioxide treatment will be administered (15 weeks of maintenance). Pts. are to continue on imatinib 800 mg/day,(or the max. tolerated dose) while receiving the arsenic trioxide. If a pt. has been taken off the arsenic trioxide, they should be continued on gleevec 800 mg per day (or the maximum tolerated dose) until there is evidence of progression of disease.

SUMMARY:
1.0 OBJECTIVES 1.1 To test the activity of arsenic trioxide in combination with imatinib in patients with CML with cytogenetic evidence of residual disease.

1.2 To determine the toxicity associated with this therapy.

DETAILED DESCRIPTION:
* Chronic myelogenous leukemia (CML) results from the clonal expansion of immature myeloid cells with the t (9,22) (Ph) translocation, that encodes the constitutively active tyrosine kinase oncogene, bcr/abl. Patients with chronic phase CML are currently being treated with either hemopoetic stem cell transplantation (HSCT), or with the recently approved tyrosine kinase inhibitor, imatinib. Previous data, using interferon in patients with CML, has shown that patients who do not achieve a major cytogenetic response (defined as >35% Ph+) have a shortened survival. These patients are often considered for HSCT. However, due to constraints of age, suitable donor, and patient choice, only a minority of patients will undergo this potentially curative procedure.
* The aim of this study is to create a uniform approach to the treatment of CML in New Mexico, with an aim of achieving complete cytogenetic response as the primary goal. A graded approach will be taken, starting out with the standard treatment (imatinib 400 mg per day), and then in patients identified as poor responders an imatinib, and arsenic combination will be offered to patients. It is hoped to find a complete cytogenetic response that exceeds the ~20% response with gleevec 800mg per day.

ELIGIBILITY:
Inclusion criteria:

* All patients, 18 years of age or older, with a diagnosis of CML.
* Patients must have a life expectancy of at least 12 weeks.
* Patients must have an ECOG performance status of 0-2.
* Patients must sign an informed consent.
* Patients should have adequate hepatic function with a total bilirubin < 2 mg/dl and SGOT or SGPT < two times the upper limit of normal, and adequate renal function as defined by a serum creatinine < 1.5 x upper limit of normal.
* Patients with CML in chronic phase on gleevec as first line therapy who fulfill the following criteria:
* Failure to achieve a complete hematologic response (CHR) after 3 months of therapy (hematologic resistance)
* Failure to achieve a complete cytogenetic response (CGCR) after > 9 months of therapy.
* Cytogenetic relapse, defined as an increase in the Ph+ cells by at least 30%.
* Hematologic relapse defined as the appearance of any of the following, confirmed by a second determination > 1 month later:

  * WBC count >20, 000,
  * Platelet count >600,000,
  * Progressive splenomegaly > 5 cm below the left intercostals margin,
  * >5% myelocytes and/or metamyelocytes in the peripheral blood,
  * Blasts or promyelocytes in the peripheral blood

Exclusion Criteria:

* Pregnant women or nursing mothers are not eligible for this trial. Patients of child bearing potential must use adequate contraception.
* Patients may receive no other concurrent chemotherapy or radiation therapy during this trial.
* Patients with severe medical problems such as uncontrolled diabetes mellitus or cardiovascular disease or active infections are not eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2004-04; Primary Completion 2005-04 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
To test the activity of arsenic trioxide in combination with imatinib in patients with CML with cytogenetic evidence of residual disease | 2 years

SECONDARY OUTCOMES:
To determine the toxicity associated with this therapy | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ian Rabinowitz, MD, Principal Investigator — University of New Mexico
Locations (2):
- United States (2):
  - University of New Mexico, Albuquerque, New Mexico
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico